CLINICAL TRIAL: NCT00056745
Title: The Role of Immunization Site in Eliciting Mucosal Immunity
Brief Title: Determining an Effective Site (Groin Versus Arm) for Giving HIV Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01AI050467 (NIH); UCLA MIG-001; R01AI050467 (NIH)
Record Dates: First submitted 2003-03-21; First posted 2003-03-24 (Estimated); Last update posted 2007-09-18 (Estimated); Status verified 2007-07

CONDITIONS: HIV Infections
Keywords: HIV seronegativity; HIV preventive vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: TBC-3B

SUMMARY:
The purpose of this study is to determine the safety and immune system response to the TBC-3B HIV vaccine when it is injected either into the groin area or into the arm. The goal is to determine which injection site is better at producing a particular type of immune response. This study is not evaluating the effectiveness of the vaccine, so volunteers must maintain low risk behavior for HIV transmission throughout the study.

DETAILED DESCRIPTION:
The goal of this vaccination study is to evaluate the safety and immunogenicity of the Therion Biologic Corporation (Cambridge, MA) TBC-3B vaccine. TBC-3B consists of live, recombinant vaccinia virus expressing the env and gag/pol genes of HIV-1 strain IIIB. TBC-3B will be administered by subcutaneous injection in the groin and in the deltoid region, with the aim of determining which site is better at inducing mucosal immune responses. Because the groin area drains to the inguinal lymph nodes, vaccines given there may stimulate local immunologic activity in the draining rectal mucosa as well as systemic immunologic activity in the blood.

Volunteers will be followed for 20 months. The first 2 months of the study will be an evaluation of volunteers' normal immune function. Volunteers will then be randomly selected to receive the TBC-3B experimental HIV vaccine in either the groin area or in the deltoid region. Neither volunteers nor study personnel will know which group the volunteer will be in until the day of the first immunization. All volunteers will receive TBC-3B.

During the 20 months of the study, volunteers will be asked to donate blood up to 14 times, undergo seven flexible sigmoidoscopies with biopsies, and receive three pairs of vaccine injections. For up to 36 days after each experimental vaccination, volunteers will be asked to abstain from activity that might spread the virus in the vaccine and put others at risk. Volunteers will receive specific instructions on how to avoid these risks. Volunteers will also be asked not to engage in receptive anal intercourse during the study.

ELIGIBILITY:
Inclusion Criteria

* HIV uninfected
* Low risk for HIV-1 (no sexually transmitted disease within 1 year of study entry, no history of injection drug use, no sex with an HIV infected individual or active injection drug user within 6 months of study entry, no unsafe sexual activity with unknown partners) or mutually monogamous relationship with a known HIV seronegative partner (per subject report) for 6 months prior to study entry
* Born after 1970
* Willingness to abstain from sexual activity for up to 30 days after each vaccination
* Willingness to abstain from receptive anal intercourse during the 20 months of the study
* Available for follow-up during the 20 month duration of the study
* Acceptable methods of contraception

Exclusion Criteria

* Immunosuppression of any type, including those related to lupus, rheumatoid arthritis, leukemia, lymphoma, generalized malignancy, agammaglobulinemia, and therapy with alkylating agents, antimetabolites, radiation, or large doses of corticosteroids
* Gastrointestinal complaints such as inflammatory bowel disease or chronic diarrhea
* Medical or psychiatric condition or occupational responsibilities which preclude volunteer's compliance with the protocol; specifically excluded are people with a history of suicide attempts, recent suicidal ideation, or who have past or present psychosis
* Prior smallpox or vaccinia-based vaccination
* Live attenuated vaccines within 60 days of study. Medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) are not exclusionary, but should be given at least 1 month prior to TBC-3B immunizations.
* Anaphylaxis or other serious adverse reactions to vaccines
* Serious allergic reaction to any substance requiring hospitalization or emergent medical care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension)
* Sexually transmitted disease in the year prior to study entry
* Genital HSV (herpes) or other ulcerative genital lesions
* Active HBV (hepatitis B) or HCV (hepatitis C) infection
* Nonprescribed injection drug use
* Pregnant or lactating women
* Acute, chronic, or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, eczema)
* Use of experimental agents within 30 days prior to study
* Household contacts with or ongoing occupational exposure to any of the following: pregnant women; children < 12 months of age; people with acute, chronic, or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, eczema); people with an immunodeficiency or using immunosuppressive medications

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12

PRIMARY OUTCOMES:
Safety of administering TBC-3B vaccinations to vaccinia naive individuals

SECONDARY OUTCOMES:
Immunogenicity of subcutaneous vaccination with 3 doses of TBC-3B administered in the groin area, as measured by increased levels of CTL activity directed to vaccinia and HIV-1 env, gag and pol gene products
immunogenicity of subcutaneous vaccination with 3 doses of TBC-3B administered in the groin area, as measured by anti-HIV-1 directed CD4+ T cell proliferative response to soluble p24 antigen
immunogenicity of subcutaneous vaccination with 3 doses of TBC-3B administered in the groin area, as measured by CD8+ T cell specificity for HIV-1 epitopes
immunogenicity of subcutaneous vaccination with 3 doses of TBC-3B administered in the groin area, as measured by serum and mucosal immunoglobulins against HIV-1 epitopes

CONTACTS AND LOCATIONS:
Overall Officials: Peter Anton, MD, Principal Investigator — University of California at Los Angeles
Locations (1):
- University of California at Los Angelos Center for HIV and Digestive Diseases, Los Angeles, California, United States